CLINICAL TRIAL: NCT05478512
Title: Front-line Venetoclax and Obinutuzumab Combination Followed by Venetoclax or Venetoclax and Zanubrutinib Combination in Patients With Residual Disease: a Minimal Residual Disease (MRD) Tailored Treatment for Young Patients With High-risk CLL
Brief Title: Front-line VenObi Combination Followed by Ven or VenZan Combination in Patients With Residual Disease: a MRD Tailored Treatment for Young Patients With High-risk CLL
Acronym: VIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL2222
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: High Risk CLL; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VenObi+Ven or VenObi+VenZan (Experimental): Patients will receive VenObi combination followed by Venetoclax single agent or Venetoclax+zanubrutinib, according to MRD.
  Interventions: Drug: VenObi+Ven or VenObi+VenZan

INTERVENTIONS:
Drug: VenObi+Ven or VenObi+VenZan — Patients will receive obinutuzumab 1000mg IV (cycle 1: day 1,8,15; Cycle2-6: day1) + venetoclax 400mg/d (preceded by a ramp-up phase) until cycle 9, day 28.
  At cycle9:
  * if uMRD = Venetoclax 400 mg/d orally until cycle 13.
  * if residual disease in the BM or PB = Venetoclax 400 mg/d + Zanubrutinib 160 mg orally twice daily until cycle 21.
  then, at cycle 21:
  * if uMRD = stop treatment
  * if residual disease in the BM or PB = zanubrutinib 160 mg orally twice daily until disease progression

SUMMARY:
Multicentric phase 2 study for previously untreated high-risk CLL patients. Patients will receive 6 courses of the Venetoclax + Obinutuzumab combination.

* Patients with stable disease or a response (CR/PR) with uMRD in the PB and BM at cycle 9 will continue treatment with Venetoclax single agent until cycle 13 and then stop treatment.
* Patients with stable disease or a response (CR/PR) with evidence of residual disease in the PB and/or BM at cycle 9 will continue treatment with Venetoclax and Zanubrutinib combination until cycle 21.

then, Patients with uMRD in the PB and BM at cycle 21 will stop treatment whereas patients with residual disease in the PB and/or BM at cycle 21 will discontinue Venetoclax and continue Zanubrutinib until disease progression.

DETAILED DESCRIPTION:
This is a multicentric phase 2 study for previously untreated high-risk CLL patients.

A. The study treatment will consist of 6 courses of the Venetoclax + Obinutuzumab combination.

B. Patients with stable disease or a response (CR/PR) with undetectable MRD (uMRD) in the PB and BM at cycle 9 will continue treatment with Venetoclax single agent until cycle 13 and then stop treatment.

C. Patients with stable disease or a response (CR/PR) with evidence of residual disease in the PB and/or BM at cycle 9 will continue treatment with Venetoclax and Zanubrutinib (VenZan) combination until cycle 21.

c1. Patients with uMRD in the PB and BM at cycle 21 will stop treatment. c2. Patients with residual disease in the PB and/or BM at cycle 21 will discontinue Venetoclax and continue Zanubrutinib until disease progression.

In all patients with uMRD, MRD will be monitored during the follow-up. Patients with a response with uMRD in the PB and BM who subsequently develop an MRD positivity will not be treated. A new treatment will start at the time of clinical disease progression according to the iwCLL criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years and 65 years or less.
2. Diagnosis of CLL meeting the iwCLL 2018 criteria.
3. Total CIRS <6, creatinine clearance >30 ml/min [Cockcroft-Gault]) and ECOG performance status of 0-1.
4. No prior treatment.
5. Patients with unmutated IGHV, and, or TP53 mutation assessed by an ERIC certified laboratory, and, or deletion 17p assessed by FISH analysis.
6. Active disease meeting at least 1 of the iwCLL 2018 criteria for treatment requirement.
7. Adequate hematologic parameters unless due to disease under study:

   * Absolute neutrophil count (ANC) ≥1.0 x 109/L unless neutropenia is clearly due to disease under study (per investigator discretion)
   * Platelet count ≥ 75,000/mm3 - OR - Platelet count ≥ 20,000/mm3 if thrombocytopenia is clearly due to disease under study (per investigator discretion)
   * Hemoglobin ≥9.0 g/dL unless anemia is clearly due to marrow involvement of CLL (per investigator discretion)
8. Adequate renal and hepatic function, per laboratory reference range at screening as follows:

   * AST/SGOT, ALT/SGPT ≤2.0 x ULN
   * Total bilirubin ≤1.5 x ULN unless considered secondary to Gilbert's syndrome, in which case ≤3 x ULN
9. QT-interval corrected according to Fridericia"s formula (QTcF) ≤450 milliseconds (ms).
10. For females of childbearing potential, a negative serum pregnancy test within 7 days of study treatment.
11. For female patients of childbearing potential, agreement to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [<1% per year] when used consistently and correctly) or remain abstinent (refrain from heterosexual intercourse) during the treatment period and to continue its use for 90 days after the last dose of zanubrutinib AND 30 days after the last dose of venetoclax AND for 18 months after the last dose of obinutuzumab (whichever date is later). For men with a female partner of childbearing potential or a pregnant female partner: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom during the treatment period and to continue its use for 90 days after the last dose of zanubrutinib, or venetoclax AND for 18 months after the last dose of obinutuzumab (whichever date is later).
12. A signed informed consent document indicating that they understand the purpose of and the procedures required for the study, including biomarkers, and are willing to participate in the study.
13. Ability and willingness to comply with the requirements of the study protocol.

Exclusion Criteria:

1. Any significant concurrent, uncontrolled medical condition or organ system dysfunction and laboratory abnormality or psychiatric disease, which, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk or prevent the subject from signing the informed consent form.
2. Known active histological transformation from CLL to an aggressive lymphoma (i.e., Richter's transformation or pro-lymphocytic leukemia);
3. known central nervous system involvement.
4. Active malignancy or systemic therapy for another malignancy within 3 years

Except:

• Malignancies surgically treated with curative intent and with no known active disease present for ≥ 3 years before randomization

* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated cervical carcinoma in situ without evidence of disease
* Surgically/adequately treated low grade, early stage localized prostate cancer without evidence of disease

  5. Co-morbidities:
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
* Any uncontrolled illness that in the opinion of the investigator would preclude administration of study therapy
* History of stroke or intracranial hemorrhage within 180 days before first dose of study drug.
* History of severe bleeding disorder or history of spontaneous bleeding requiring blood transfusion or other medical intervention due to thrombocytopenia or inherited or acquired bleeding disorders due to deficiency or functional abnormality of any coagulation proteins.
* History of significant cardiovascular disease, defined as:

  1. Congestive heart failure greater than New York Heart Association (NYHA) class II according to the NYHA functional classification.
  2. Unstable angina or myocardial infarction with 6 months of enrollment.
  3. Serious cardiac arrhythmia or clinically significant ECG abnormality: corrected QT wave (QTcF) > 480 msec based on the Fridericia's formula or other ECG abnormalities including second-degree atrioventricular block type II, third-degree atrioventricular block. Participants who have a pacemaker will be allowed on study despite ECG abnormalities or the inability to calculate the QTc.
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1, Day 1
* History of tuberculosis within the last five years or recent exposure to tuberculosis equal to or less than 6 months.
* History of progressive multifocal leukoencephalopathy (PML)
* History of HIV infection or active hepatitis B (chronic or acute) or hepatitis C infection 1. Patients with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV DNA is undetectable. These patients must be willing to take appropriate anti-viral prophylaxis as indicated and undergo monthly DNA testing.

  2. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Inadequate renal function: CrCl < 30 mL/min.
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Known intolerance or hypersensitivity to any of the components of the therapeutic regimen
* Receipt of live-virus vaccines within 28 days prior to the initiation of study treatment or need for live-virus vaccines at any time during study treatment.
* Prior major surgical procedure within 4 weeks of study, or anticipation of need for a major surgical procedure during the course of the study
* Known condition or other clinical situation that would affect oral absorption.
* Psychiatric illness/social situations that would interfere with study compliance.
* Inability to swallow a large number of tablets.

  6. Concomitant medications and drug interactions:
* Patients who are on treatment with the following agents within 7 days prior to treatment:

Strong CYP3A inhibitors such as fluconazole, ketoconazole, and clarithromycin Strong CYP3A inducers such as rifampin, carbamazepine and strong inhibitors or inducers of CYP2C8, CYP2C9 and CYP2C19. The same applied for moderate inhibitors or inducers of CYP3A Requires warfarin, marcumar, or phenprocoumon (due to potential drug-drug interactions that may potentially increase the exposure of warfarin or phenprocoumon)

• Prior anti-CD20 monoclonal antibody therapy for non-malignant indication

7. Females who are currently pregnant or breastfeeding.

8. Participation in a separate investigational therapeutic study unless authorized by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Front-line VenObi efficacy in terms of MRD negativity | at month 9
  Evaluation of front-line treatment (VenObi) efficacy in terms of percentage of patients who achieve Undetectable Minimal Residual Disease at the end of combination therapy
VenZan efficacy in terms of MRD negativity | at month 21
  Evaluation of treatment (VenZan) efficacy in terms of percentage of patients who achieve Undetectable Minimal Residual Disease in patients with residual disease at the end of combination therapy with VenObi

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - Ematologia AOU Careggi, Florence
  - Ematologia IRST D.Amadori, Meldola
  - Ematologia AO di Perugia, Perugia
  - Ematologia Ospedale S.M. delle Croci, Ravenna
  - Ematologia Ospedale Infermi, Rimini
  - Ematologia Policlinico Gemelli, Roma
  - Ematologia Policlinico Umberto I, Roma
  - Ematologia AOUS - Policlinico S. M. alle Scotte, Siena